CLINICAL TRIAL: NCT05793502
Title: Study on Effectiveness and Safety of LBBaP With Solia S and Selectra 3D Developed by BIOTRONIK
Status: Recruiting | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Chen Keping, Clinical Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 20230320
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Consented to Participate in the Trial and Signed an ICF; Patients With an Indication for PM Implantation or CRTP

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Permanent pacemaker implantation or cardiac resynchronization therapy: Patients with an indication for permanent pacemaker implantation or CRT
  Interventions: Device: Solia S and Selectra 3D Developed by BIOTRONIK

INTERVENTIONS:
Device: Solia S and Selectra 3D Developed by BIOTRONIK — LBBaP with Solia S and Selectra 3D Developed by BIOTRONIK

SUMMARY:
This study is aimed to assess the effectiveness and safety of LBBaP with Solia S and Selectra 3D in the Chinese population by analyzing the operation success rate and the system stability during follow-up visits.

DETAILED DESCRIPTION:
Traditional ventricular pacing leads are placed in and around the right ventricular apex (RVA), which are easy to operate. The long-term safety and efficacy of right ventricular pacing (RVP) in the treatment of bradycardia arrhythmia have been demonstrated. However, it is shown by CTOPP (Canadian Trial of Physiologic Pacing) study (1), MOST (Micro-Optical Sectioning Tomography) study (2) and UKPACE (United Kingdom Pacing and Cardiovascular Events) study (3) that long-term and high-proportion right ventricular apical pacing (RVAP) may lead to ventricular systolic asynchrony, and accordingly increase the risks of cardiac failure (cardiac insufficiency) and atrial fibrillation (AF).

The concept of His bundle pacing (HBP) has been put forward for a long time, in which His bundle is directly stimulated to synchronously excite the ventricles mainly through the conduction of the His-Purkinje system (HPS) in the electrical activity of the heart. The study performed by Vijayaman et al. (4) shows that HBP can reduce the long-term mortality and the risks of hospitalization for cardiac failure and upgrading to CRT compared with the traditional RVAP. However, HBP surgery has the following disadvantages: (1) It is rather difficult to fix the leads, the operation duration is long, the suture removal duration is long, and the learning curve of doctors is long; (2) The threshold value is high during implantation and may further increase in the long term, and the sensory power is rather low. Therefore, the implantation of spare leads is recommended in relevant guidelines, increasing the hardware burden in patients; (3) The implantation site of patients with conduction block below His bundle is rather difficult or unable to cross the block site.

In order to improve the HBP surgery, Chinese doctors have put forward LBBaP in recent years, arousing widespread concern all over the world. Dedicated sheath tubes and electrode leads are adopted in the technique. Specifically, electrode leads are "screwed" into the left bundle branch area under the left ventricular intima from the right ventricular septum (RVS), and the left bundle branch pacing (LBBP) is performed to improve bradycardia. Compared with HBP, LBBP has the following advantages: (1) As the implantation site is easier to locate, the operation difficulty is reduced; (2) With a lower and more stable threshold, the sensitivity is better; (3) Distal block is corrected; (4) An enough space is left for atrioventricular junction ablation.

At present, it is collectively known as HBP in the international community. LBBaP refers to conduction system pacing, the performing of which depends on dedicated tools or instruments. In early times, the positioning and fixation of shaping steel wires in combination with active-fixation leads adopted in the technique were realized with the aid of a mapping catheter. The operation success rate of HBP was rather low and LBBaP could not be realized. With the introduction of dedicated sheath tubes by various manufacturers, the operation success rate has been greatly improved. However, there are no enough data derived from large-scale studies at home and abroad on the effectiveness and safety of LBBaP with Selectra 3D and Solia S developed by BIOTRONIK at present.

This study is aimed to assess the effectiveness and safety of LBBaP with Solia S and Selectra 3D in the Chinese population by analyzing the operation success rate and the system stability during follow-up visits.

ELIGIBILITY:
Inclusion criteria

1. All patients for whom it is the first time to receive permanent pacemaker implantation or CRT, and on whom LBBaP will be performed for trial.
2. Willingness to participate in the investigation and sign the ICF
3. Ability and willingness to perform all follow-up visits at the investigation sites

Exclusion criteria

1. Age less than 18 years
2. Patients with cardiac amyloidosis
3. Patients with ventricular hypertrophy (interventricular septum diastolic thickness measured from two-dimensional echocardiography: ≥ 15 mm; or, interventricular septum diastolic thickness for patients with a definite family history: ≥ 13 mm)
4. Participating in other intervention clinical trials
5. Life-expectancy less than one year
6. Pregnancy and/or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for permanent pacemaker implantation or CRT
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
Implantation success rate of LBBaP | During the surgery
  Implantation success rate of LBBaP
Intraoperatively, the incidence of serious adverse events for devices associated with Solia S and Selectra 3D implantation rate | During the surgery
  Intraoperatively, the incidence of serious adverse events for devices associated with Solia S and Selectra 3D implantation rate
Occurrence of serious adverse events rate | From the time of surgery to the 12-month post-implantation visit
  The incidence of serious adverse events associated with permanent pacemaker implantation or cardiac resynchronization from the time of surgery to the 12-month post-implantation visit Incidence of serious adverse events associated with the treatment procedure

SECONDARY OUTCOMES:
Number of participants with abnormal pacing parameters and abnormal ECG readings | 1 month and 12 months post-procedure
  Assessment of the consistency of pacing parameters and ECG characteristics at 1 month and 12 months postoperatively
Changes of cardiac ultrasound values (including LVEF, LVESD and LVEDD) | 12 months post-procedure.
  At the 12-month follow-up, a cardiac ultrasound was performed, and the primary measurements included LVEF, LVESD, and LVEDD, comparing changes in LVEF, LVESD, and LVEDD at the 12-month follow-up with those prior to hospital discharge
Changes of NYHA class | 1 month and 12 months post-procedure
  The extent of change in NYHA classification and number of subjects at 1 and 12 months postoperatively.
Changes of EQ-5D-5L assessment | 1 month and 12 months post-procedure
  Extent of change in EQ-5D-5L assessment at 1 and 12 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Chen Keping, Doctor, Principal Investigator — Fu Wai Hospital, Chinese Academy of Medical Sciences, Fu Wai, China
Locations (1):
- Shanxi Cardiovascular Hospital, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No
The project is a prospective, multicenter and single-group observational study. A total of 1,000 subjects will be enrolled at 20 investigation sites within the territory of China. All subjects enrolled will receive permanent pacemaker implantation or cardiac resynchronization therapy (CRT), and LBBaP will also be performed on them for trial. They will be followed up at pre-hospital discharge, and 1 month and 12 months post-procedure. Data collected in the investigation will be analyzed to assess the effectiveness and safety of LBBaP with Solia S and Selectra 3D in the Chinese population.